CLINICAL TRIAL: NCT03912896
Title: Taekwondo for Children With Autism Spectrum Disorder: The Impact on Social Interaction Skills in Everyday Life
Brief Title: Taekwondo for Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Julie Kugel, Associate Professor, OTD Program Director, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 5180418
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Autism Spectrum Disorder
Keywords: taekwondo; Autism Spectrum Disorder; occupational therapy; Social interaction skills; child participants
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Children with autism spectrum disorder (Experimental)
  Interventions: Behavioral: Taekwondo

INTERVENTIONS:
Behavioral: Taekwondo — Children will participate in a 7-week taekwondo program.

SUMMARY:
This study uses a mixed methods design to understand the effectiveness of using taekwondo as an intervention for children with ASD and its effect on social interaction skills and everyday life. Qualitative research emphasizes that meaning can be explained and interpreted only by those who experience it. A pretest-posttest design will be used to describe what occurs after the introduction of the taekwondo intervention and understand the changes that occur after exposure. Collecting information through the lived experiences and observations from the parents will be collated with the pre and post results of the children participants' social interaction skills.

Qualitative data will be collected through pre and post semi-structured interviews with the parents to understand their observations of their child before and after completing the taekwondo program. Interviews will also be conducted with the child to understand their perspectives on physical activity participation. Interview questions will also explore how the effectiveness of the program has impacted the children's engagement in daily activities.

Quantitative research will be collected through pre and post results from the Autism Social Skills Profile-2 ([ASSP] assessment that will be completed by the parents. The ASSP-2 provides a comprehensive measure of social functioning for children and adolescents with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Formal diagnosis of autism spectrum disorder (ASD)
* Able to follow and understand English verbal instructions during the screening process.
* No experience or prior experience with martial arts.
* Able to walk and move without using adaptive equipment

Exclusion Criteria:

* Physical disabilities that would prevent participation in taekwondo (e.g. wheelchair bound)

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Subject response to taekwondo | Change between baseline and week 7.
  Autism Social Skills Profile-2 (ASSP-2) will be administered at baseline prior to taekwondo instruction and then administered again at week 7. The ASSP-2 has 49 items and each are rated on a 4-point Likert scale with a minimum score of 1 representing never and a maximum score 4 representing very often for each item. This is a composite measurement. The scale ranges from a total raw score of 49 to a maximum of 196. There are three subscales: 20 social/emotional reciprocity (SER) items, 11 structured play activity (SPA) items, and 11 detrimental social behaviors (DSB) items. One component skill is measured as both an SER and SPA subscale. Standard scores have a mean of 100 and a standard deviation of 15. The higher the scores for each section means that the child does not have difficulties with social skills for that subscale. The lower the scores shows a deficit in each area.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Kugel, Principal Investigator — Loma Linda University Health
Locations (1):
- Loma LInda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No